CLINICAL TRIAL: NCT02885623
Title: Clinical Significance of CX3CR1 Adhesion Molecule-expressing Myeloid and Lymphoid Cells in Hematologic Malignancy
Brief Title: Role of CX3CR1-expressing Cells in Hematologic Malignancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Saint Vincent's Hospital, Korea (Other)
Responsible Party: Principal Investigator, Jeong-A Kim, Professor, Division of Hematology, Department of Internal Medicine, Saint Vincent's Hospital, Korea
Other Study IDs: 001
Record Dates: First submitted 2016-08-23; First posted 2016-08-31 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: CX3CR1 Protein; Diffuse Large B Cell Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the clinical significance of CX3CR1-expressing myeloid and lymphoid cells in patients of hematologic malignancy.

Tumor cells either express membrane molecules or release tumor-derived soluble factors able to alter myelopoiesis and lymphopoiesis. Myeloid cells expressing CD11b play a critical role in sustaining cancer progression. Also, the fractalkine (CX3CL1; Fkn)/CX3CR1 axis plays an important function in the pathophysiology of various forms of cancers. Fkn is the only known ligand for CX3CR1, and it triggers recruitment of CX3CR1-positive cells through its unique receptor, CX3CR1. Therefore, the investigators focused the prognostic significance of CD11b+ myelo-monocytic cells expressing CX3CR1 and CD3+ lymphoid cells expressing CX3CR1 in the clinical outcomes of newly diagnosed Diffuse Large B-cell Lymphoma (DLBCL) and Multiple myeloma (MM).

DETAILED DESCRIPTION:
Bone marrow aspirates will be obtained from newly diagnosed MM and DLBCL patients at the time of diagnosis and relapse. Peripheral blood will be obtained at the time of diagnosis, finishing treatment, 3 months after treatment and relapse.

The investigators will analyze the cell fractions of CD11b+ CX3CR1+ cells and CD3+CX3CR1+ cells in blood samples by flowcytometry. The investigators will find out the relationship between the tested cells and clinical outcome in MM and DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Subject newly diagnosed multiple myeloma.
* Subject newly diagnosed diffuse large B cell lymphoma.

Exclusion Criteria:

* History of other hematologic malignancy
* History of previous chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed multiple myeloma patients newly diagnosed diffuse large B cell lymphoma patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
Death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-A Kim, MD, Ph.D, Principal Investigator — Saint Vincent's Hospital, Korea
Locations (1):
- The Catholic University of Korea, St.Vincent's hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided